CLINICAL TRIAL: NCT02331316
Title: Drinking Water To Prevent or Reduce Weight Gain - An Online Randomized Controlled Trial With Adult Participants
Brief Title: Drinking Water to Reach or Maintain a Healthier Weight
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: PI Retired study unfunded
Sponsor: ThinkWell (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: ThinkWell PLOT-02
Record Dates: First submitted 2015-01-01; First posted 2015-01-06 (Estimated); Last update posted 2021-03-23 (Actual); Status verified 2021-03

CONDITIONS: Obesity; Dietary Modification
Keywords: obesity; diet; weight; hunger; public led trial
MeSH Terms: conditions — Obesity; Body Weight

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Daily extra water intake 2L (Experimental): Timing of daily extra water intake
  intervention-A: extra water intake: 8 8oz glasses of water a day (2L) - 2 first thing in the morning before breakfast, 2 before midday or midday meal, 2 before afternoon meal and 2 before evening meal.
  Intervention-B: Drink extra water at anytime over 24 hours
  Interventions: Other: Daily extra water intake
- Daily extra water intake 1L (Experimental): Timing of daily extra water intake
  Intervention-A: 4 8oz glasses of water a day (1L) - 1 first thing in the morning before breakfast, 1 before midday or midday meal, 1 before afternoon meal and 1 before evening meal.
  Intervention-B: Drink extra water at anytime over 24 hours
  Interventions: Other: Daily extra water intake
- Daily extra water intake 500ml (Experimental): Timing of daily extra water intake
  Intervention-A: 2 8oz glasses of water a day (500ml) - each half an hour before a meals.
  Intervention-B: Drink extra water at anytime over 24 hours
  Interventions: Other: Daily extra water intake
- Daily extra water intake 120ml (Experimental): Timing of daily extra water intake
  Intervention-A: 1/2 a glass of water on waking (120ml). If you forget to drink your water first thing, do not drink it later in the day, just skip this day and drink ½ a glass the next day on waking.
  Intervention-B: Drink extra water at anytime over 24 hours
  Interventions: Other: Daily extra water intake

INTERVENTIONS:
Other: Daily extra water intake — Intervention-A: Timing of assigned daily extra water intake specified
  Intervention-B: Daily extra water assigned at any time during 24 hour period

SUMMARY:
The purpose of this study is to find out if drinking extra water helps people lose or maintain weight loss and reduce hunger and, if so, what volume of water is most effective and when is it best to drink it.

DETAILED DESCRIPTION:
Obesity is a major public health problem. Observational data suggest that drinking water is associated with a healthier weight. Indeed advice to drink extra water to help with weight control is widespread (eight 8oz glasses or 2L of water a day is a common recommendation). The public spends billions of dollars on bottled water in the belief that it works and people are increasingly carrying water with them throughout the day. However, a systematic review of randomized controlled trials looking at the effectiveness of drinking extra water to help reduce weight or weight gain or produce changes in surrogate markers such as appetite or caloric intake undertaken by our group showed that currently there is an absence of reliable evidence to support the recommendation to drink water.

It is important to establish whether drinking extra water is indeed helpful for weight control and, if so, what is the optimal quantity to recommend, as this could have an important impact of public health and public health policies if it is indeed effective. Tap water is so readily available in this country that even if the improvement in weight maintenance or reduction is small, this will be a cost-effective intervention. If it is not effective, then it is important that people know this so that they can make an informed choice about buying bottles of water for their health.

The primary clinical question the study will address is does drinking extra water prevent or reduce weight gain?

The secondary clinical questions it will ask are:

1. Does drinking water reduce hunger or increase satiety
2. Does drinking water increase participants' sense of well-being
3. What is the effect of the different volumes of water on nocturnal urination patterns?

Once participants decide to take part in this trial, they will be asked to drink a specific amount of water at particular times of the day for 6 months. A computer will decide by chance the amount of water they will be asked to drink each day of the trial and the times at which to drink this.

There are different amounts and different times that people will be asked to drink water, this is so that investigators can find out if there is an optimal volume of water to drink, and a best time to drink water to reduce headaches or hunger. The least amount of water the computer could ask participants to drink is half a glass (that is 4oz or 120ml). The largest volume of water the computer could ask a participant to drink would be eight glasses of water a day (a total of 64oz or 2L) spread across the day (that is not all at once). Once the computer has assigned participants to a particular volume and times to drink water, these will remain the same for every day throughout the study.

Participant will be asked to provide some brief information about themselves at the beginning of the study (for example, age, sex, height and whether they exercise, smoke or not). During the study they will be asked to weigh themselves and record this, their dietary habits and the amount they drink will be stored on a private and confidential page on the study website. They will be asked to fill in [2] confidential short surveys about how they feel and their views, one at the start and one at the end of the study

ELIGIBILITY:
Inclusion Criteria:

* Any adult (defined as someone aged 18 or above) for who advice to drink extra water is not contraindicated.

Exclusion Criteria:

General:

1. < 18 years of age
2. No personal email address
3. Pregnancy
4. Ecstasy recreational drug use

Health conditions:

1. Impaired renal function
2. Chronic bowel problems
3. Low sodium levels
4. Diabetes insipidus
5. Schizophrenia or history of psychosis
6. Congestive heart failure
7. Current chemotherapy treatment
8. Anorexia
9. bulimia

Concurrent Medications:

1. Taking regular non-steroidal anti-inflammatory drugs
2. Diuretics (e.g. thiazides, indapamide, loop diuretics), also called "water tablets"
3. Anti-depressants Selective serotonin re-uptake inhibitors (SSRIs), Tricyclic and tetracyclic antidepressants (TCAs),monoamine oxidase inhibitor (MAOIs)
4. Anti-psychotics (e.g. haloperidol)
5. Anti-convulsants (e.g. sodium valproate, carbamazepine)

Implicit exclusions:

1. People without internet access
2. People who cannot read 3 People without the ability to understand the website and informed consent documents

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-01 (Estimated); Primary Completion 2019-08 (Estimated); Study Completion 2019-11 (Estimated)

PRIMARY OUTCOMES:
Weight loss or maintenance recorded online using participant reported outcome measures(PROMS) | 6 months
  Weight loss or maintenance recorded online using participant reported outcome measures(PROMS). Participants will be asked to record weight using a supplied body mass index calculator and home weight scales weekly or as a minimum at baseline and close of study

SECONDARY OUTCOMES:
Hunger intensity and satiety recorded online using participant reported outcome measures(PROMS) | 6 months
  Hunger intensity and satiety recorded online using participant reported outcome measures(PROMS). Participants will be asked to self report hunger and satiety levels using a mobile app, web or journal using a visual analog scale (VAS ) on a daily basis or as a minimum at baseline and close of study
Well-being as measured by The PROMIS Well-being measure | 6 months
  The PROMIS Well-being measure will be administered to participants monthly,
  There will be a VAS Mood scale where they can record sad to happy mood at the same time they record hunger
Nightly micturition frequency as measured by self report | 6 months
  Participants will self report weekly if nightly micturition frequency increases, decreases or there is no change

CONTACTS AND LOCATIONS:
Overall Officials: Amanda J Burls, MD, Principal Investigator — ThinkWell and City University London; Martin Cartwright, PhD, Principal Investigator — City, University of London
Locations (1):
- ThinkWell and City University London, Oxford, Oxfordshire, United Kingdom

REFERENCES:
- [Background] 1 Price A, Burls A, Spurden D, et al. Water intake for weight reduction: a Systematic Review. PROSPERO. 2013.http://www.crd.york.ac.uk/PROSPERO/display_record.asp?ID=CRD42013004998
- [Background] 1 Price A, Burls A. PLOT-IT Public Led Online Trials Infrastructure and Tools. In: Force 2015. Oxford UK: : Force2015 2015. doi:DOI: 10.13140/2.1.1992.6082